CLINICAL TRIAL: NCT01910857
Title: Improving Hypertension Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Progressive Community Health Center (Unknown)
Responsible Party: Principal Investigator, Theodore Kotchen, MD, Professor Emeritus, Assoc Dean for Clinical Research, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO16801; HWPP (Other Grant/Funding Number: 2011D-41)
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Lifestyle counseling. 6 group meetings,facilitated by community health worker, focusing on lifestyle change, eg, weight loss, physical activity, low salt, stress reduction
  Interventions: Behavioral: Lifestyle counseling
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Lifestyle counseling — weight reduction, low salt, physical activity, stress reduction
  Arms: Lifestyle counseling

SUMMARY:
* The overall hypothesis for the project is that racial health disparities will be reduced by improving hypertension control in African Americans.
* This will be accomplished through the development, implementation, and evaluation of a cost-effective hypertension control strategy based on the involvement of a community health worker.

ELIGIBILITY:
Inclusion Criteria:

* African Americans with uncontrolled hypertension, followed at Progressive Community Health Centers

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure (mmHg) | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lisbon Avenue Health Center, Milwaukee, Wisconsin
  - Hillside Family Health Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Tully M, Kos A, Eastwood D, Kusch J, Kotchen T. Implementation of an Adjunct Strategy to Reduce Blood Pressure in Blacks with Uncontrolled Hypertension: a Pilot Project. Ethn Dis. 2015 Spring;25(2):168-74. PMID 26118144